CLINICAL TRIAL: NCT03855800
Title: Molecular Detection of Advanced Neoplasia in Pancreatic Cysts (IN-CYST)
Brief Title: Molecular Detection of Advanced Neoplasia in Pancreatic Cysts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-008436; 2U01CA210138 (NIH)
Record Dates: First submitted 2019-01-31; First posted 2019-02-27 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Pancreas Cyst
MeSH Terms: conditions — Pancreatic Cyst | interventions — Blood Specimen Collection; Defecation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinical Follow-up (Experimental): Participants not undergoing surgery will be assigned to the "Clinical Follow-up" study group. Blood, stool, pancreatic juice and cyst fluid collection will be done as per protocol. All participants in the Clinical Follow-up group will be contacted yearly for a telephone interview until they undergo surgery, die, receive a diagnosis that excludes them from the study, or for 5 years, and interval medical records will be obtained and reviewed. During follow-up results of clinically indicated follow-up imaging studies will be abstracted
  Interventions: Diagnostic Test: Blood, stool, pancreatic juice and cyst fluid collection; Procedure: Endoscopy Exam
- Surgical (Other): Participants scheduled for surgical resection after their initial clinical evaluation will be assigned to the "Immediate Surgery" study group. Blood, stool, pancreatic juice and cyst fluid collection will be done as per protocol. Participants in the Immediate Surgery group will be followed until the surgical pathology of their pancreatic cyst is known.
  Interventions: Diagnostic Test: Blood, stool, pancreatic juice and cyst fluid collection; Procedure: Pancreatic Surgery

INTERVENTIONS:
Diagnostic Test: Blood, stool, pancreatic juice and cyst fluid collection — Blood and stool will be collected at baseline from all study participants. Those in the Immediate Surgery group may undergo endoscopic pancreatic juice collection before surgery, either at the time of a clinically indicated endoscopic ultrasound (EUS) exam or during an optional pre-operative research endoscopy. Pancreatic cyst fluid will also be obtained from all participants in the Immediate Surgery group, either at the time of surgery, or during a clinically indicated preoperative EUS FNA procedure, or both. Pancreatic juice and cyst fluid will be collected opportunistically from participants in the Clinical Follow-up group who undergo a clinically indicated EUS, EUS FNA, or endoscopy exam.
Procedure: Pancreatic Surgery — Surgical resection of pancreatic cyst
  Arms: Surgical
Procedure: Endoscopy Exam — Clinically indicated endoscopic ultrasound
  Arms: Clinical Follow-up

SUMMARY:
Researchers are trying to find out whether new tests ("biomarkers") of blood, stool, pancreas cyst fluid, or pancreas juice can be used to diagnose malignant or pre-malignant changes in pancreas cysts.

DETAILED DESCRIPTION:
Subjects with Fukuoka Worrisome (FW) or Fukuoka High Risk (FHR) pancreatic cysts will be enrolled and assigned to Immediate Surgery or Clinical Follow-up groups based on clinical management as determined by the treating physicians. Blood, stool, pancreas cyst fluid, and pancreas juice specimens will be collected from participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pancreatic cystic lesions meeting Fukuoka worrisome or Fukuoka high-risk criteris
* Patients with suspected cystic neoplasm of the pancreas
* Able to provide written informed consent

Exclusion Criteria:

* Pregnant and/or nursing
* Incarceration
* Imaging showing possible pancreatic cancer
* Prior history of pancreatic cancer or pancreatic surgery
* History of receiving systemic chemotherapy or abdominal radiation within the last 5 years
* Previous therapy for a pancreatic cystic lesion
* History of pancreatic necrosis
* Diagnosis of cancer (other than non-melanoma skin cancer) within the last 5 years

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2018-05-11 (Actual); Primary Completion 2030-12-30 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
Biospecimen Acquisition | 5 years
  Number of biospecimens collected
High grade dysplasia (HGD) or cancer diagnosis in Immediate Surgery group | 5 years
  To validate the diagnostic accuracy of cyst fluid methylated DNA marker (MDM) assays for detection of HGD and cancer in pancreatic cysts undergoing surgical resection

SECONDARY OUTCOMES:
High grade dysplasia (HGD) or cancer diagnosis in clinical follow up group | 5 years
  To evaluate the performance of cyst fluid MDM assays for predicting development of HGD or cancer during 3-year follow-up in study patients who are initially managed non-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Shounak Majumder, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials